CLINICAL TRIAL: NCT04005157
Title: A Multi-center Study of Electromagnetic Navigation Bronchoscopy (ENB) Guided Microwave Ablation for Early-stage Peripheral Lung Cancer
Brief Title: ENB Guided MWA for Early-stage Peripheral Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017YFC0112702-MWA
Record Dates: First submitted 2019-06-20; First posted 2019-07-02 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
Keywords: Electromagnetic navigation bronchoscopy(ENB); Microwave ablation; Peripheral lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing bronchoscopic MWA (Experimental): Patients meeting the inclusion criteria will be enrolled in the study and undergo ENB guided MWA. Chest CT will be performed at 1 day after the procedure to confirm the complications and then at 1 month, every 3 months for 2 years, and every 6 months for 3 years thereafter after the procedure. PET/CT will be performed 3 months after MWA to assess the treatment response.
  Interventions: Procedure: MWA; Device: ENB

INTERVENTIONS:
Procedure: MWA — Patients diagnosed with early-stage NSCLC and signing the informed consent will undergo MWA with the guidance of ENB.
Device: ENB — ENB (LungCare Medical Technologies Ltd., Inc, Suzhou, China)will be used to guide bronchoscope into the accurate location of the lesion during MWA.

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of electromagnetic navigation bronchoscopy (ENB) guided microwave ablation (MWA) for the treatment of early-stage peripheral lung cancer.

DETAILED DESCRIPTION:
The study is designed as a multi-center prospective trial with one arm. There will be 5 centers participating the study. Patients diagnosed with early-stage non-small cell lung cancer (NSCLC) that are nonsurgical candidate will be enrolled in the study. Sixty patients are expected to be enrolled in the study. The purpose of the study is to evaluate the efficacy and safety of ENB guided MWA for the treatment of patients with early-stage nonsurgical NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral lung nodules demonstrated to be NSCLC by pathology with the clinical stage of IA.
2. The length-diameter of the tumors are more than 8 mm and no more than 30 mm.
3. Patients are unsuitable for surgery assessed by multi-modality treatment and agree to the primary treatment of ablation.
4. Patients have good compliance and sign the informed consent.

Exclusion Criteria:

1. Patients cannot receive bronchoscopy for the severe cardiopulmonary dysfunction and other indications.
2. Patients have contraindications of general anesthesia.
3. Chest CT suggests that navigation bronchoscopy technology cannot guide treatment equipment to reach the peripheral lung lesion.
4. Chest CT or bronchoscopy shows that the bronchial lumen occlusion or deformation leading to the guided and treatment equipment cannot reach the peripheral lung lesion.
5. There are large blood vessels or important structures adjacent to peripheral lung lesion.
6. Researchers consider the patient do not fit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | Three months after ablation
  Tumor response will be evaluated at 3 months after ablation. Objective response rate（ORR） is the proportion of patients with complete responses and partial responses according to the modified RECIST criteria.

SECONDARY OUTCOMES:
Arrival rate of the locatable wire | During the procedure
  Disease progression is evaluated based on the changes of the tumor on computed The arrival rate is the proportion of the locatable wire reaching the location of the tumor accurately.
Progression-free survival (PFS) | At least 3 months
  Disease progression is evaluated based on the changes of the tumor on computed tomography (CT) and/or positron emission tomography/computed tomography (PET/CT) according to modified RECIST criteria.
Overall survival (OS) | From the time of treatment to the time of the patient death with a follow-up period of 5 years
  Overall survival（OS) is evaluated after the treatment of ablation until the patient death.
Complication rate | From the time of treatment to one month after ablation
  Complications refer to serious operation-related adverse events during and after the operation, such as pneumothorax, bleeding and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie F, Zheng X, Xiao B, Han B, Herth FJF, Sun J. Navigation Bronchoscopy-Guided Radiofrequency Ablation for Nonsurgical Peripheral Pulmonary Tumors. Respiration. 2017;94(3):293-298. doi: 10.1159/000477764. Epub 2017 Jul 6. PMID 28683443
- [Background] Yang X, Ye X, Zheng A, Huang G, Ni X, Wang J, Han X, Li W, Wei Z. Percutaneous microwave ablation of stage I medically inoperable non-small cell lung cancer: clinical evaluation of 47 cases. J Surg Oncol. 2014 Nov;110(6):758-63. doi: 10.1002/jso.23701. Epub 2014 Jun 25. PMID 24965604
- [Background] Koizumi T, Tsushima K, Tanabe T, Agatsuma T, Yokoyama T, Ito M, Kanda S, Kobayashi T, Yasuo M. Bronchoscopy-Guided Cooled Radiofrequency Ablation as a Novel Intervention Therapy for Peripheral Lung Cancer. Respiration. 2015;90(1):47-55. doi: 10.1159/000430825. Epub 2015 May 30. PMID 26044954
- [Background] Liu H, Steinke K. High-powered percutaneous microwave ablation of stage I medically inoperable non-small cell lung cancer: a preliminary study. J Med Imaging Radiat Oncol. 2013 Aug;57(4):466-74. doi: 10.1111/1754-9485.12068. Epub 2013 May 8. PMID 23870347
- [Background] Sonntag PD, Hinshaw JL, Lubner MG, Brace CL, Lee FT Jr. Thermal ablation of lung tumors. Surg Oncol Clin N Am. 2011 Apr;20(2):369-87, ix. doi: 10.1016/j.soc.2010.11.008. PMID 21377589